CLINICAL TRIAL: NCT02254343
Title: Effects of Proximal and Distal Robot-assisted Therapy Combined With Functional Training on Stroke Rehabilitation
Brief Title: Effects of Proximal and Distal Robot-assisted Therapy Combined With Functional Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 103-3564A3
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Stroke
Keywords: stroke rehabilitation; robot-assisted therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- proximal robot-assisted therapy (Experimental): treatment programs will target to shoulder and elbow portions of upper extremity via the InMotion2 robotic system
  Interventions: Device: proximal robot-assisted therapy
- distal robot-assisted therapy (Experimental): the InMotion3 robot system will be used to execute treatment programs focus on wrist movements. It includes three degrees of freedom to allow wrist flexion/extension, abduction/adduction, and pronation/supination.
  Interventions: Device: distal robot-assisted therapy
- individualized intensive therapy (Active Comparator): individualized occupational therapy which is dose-match to robot-assisted therapy, based on task-oriented principle.
  Interventions: Behavioral: individualized intensive therapy

INTERVENTIONS:
Device: proximal robot-assisted therapy
  Arms: proximal robot-assisted therapy
Device: distal robot-assisted therapy
  Arms: distal robot-assisted therapy
Behavioral: individualized intensive therapy
  Arms: individualized intensive therapy

SUMMARY:
The purpose of this study is to compare the training effects of robot-assisted therapy focus on proximal part, distal part, or total segment of upper extremity, respectively.

ELIGIBILITY:
Inclusion Criteria:

* unilateral stroke that verified by CT scan
* Time since stroke more than 6 months
* moderate and mild upper limb motor impairment identified from the UE subtest of FMA range from 10 to 50
* Mini-Mental State Examination (MMSE) more than 24 points is needed to follow commands

Exclusion Criteria:

* serious visual or visual perception problems
* orthopedic or other neurological problems occurred in recent 6 months
* attend any other study in recent 3 months

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change scores of Fugl-Meyer assessment(FMA) | baseline, 2 weeks, 4 weeks

SECONDARY OUTCOMES:
Change scores of Box and block test (BBT) | baseline, 2 weeks, 4 weeks
Change scores of Action research arm test (ARAT) | baseline, 2 weeks, 4 weeks
Change scores of Medical Research Council scale (MRC) | baseline, 2 weeks, 4 weeks
Change scores of Modified Ashworth scale (MAS) | baseline, 2 weeks, 4 weeks
Change scores of Myoton | baseline, 4 weeks
Change scores of Wolf Motor Function Test (WMFT) | baseline, 2 weeks, 4 weeks
Change scores of Chedoke Arm and Hand Activity Inventory (CAHAI) | baseline, 4 weeks
Change scores of Functional independent measure (FIM) | baseline, 2 weeks, 4 weeks
Change scores of Stroke Impact Scale (SIS 3.0 version) | baseline, 2 weeks, 4 weeks
Change scores of EuroQol Quality of Life Scale (EQ-5D) | baseline, 4 weeks
Change scores of Hand strength | baseline, 2 weeks, 4 weeks
Change scores of Motor activity log (MAL) | baseline, 4 weeks
Change scores of ABILHAND Questionnaire | baseline, 4 weeks
Change scores of 10-meter walking test | baseline, 4 weeks
Change scores of Nottingham Extended ADL Questionnaire (NEADL) | baseline, 4 weeks
Change scores of Adelaide Activities Profile (AAP) | baseline, 4 weeks
Change scores of Montreal Cognitive Assessment (MoCA) | baseline, 4 weeks
Change scores of Number stroop test | baseline, 4 weeks
Change scores of Accelerometer | baseline, 4 weeks
Change scores of Revised Nottingham Sensory Assessment (rNSA) | baseline, 4 weeks
Change scores of Algometer | baseline, 4 weeks
Change scores of kinematic analysis | baseline, 4 weeks
Change scores of Adverse effects | baseline, 2 weeks, 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yi Wu, ScD, Principal Investigator — Chang Gung Memorial Hospital
Locations (2):
- Taiwan (2):
  - Chang Gung Memorial Hospital, Kwei-Shan, Tao-Yuan
  - Lo-Sheng Sanatorium and Hospital, Kwei-shan, Toayuan County